CLINICAL TRIAL: NCT02286427
Title: A Comparative Study of the Healing of Chronic Skin Ulcers of Recessive Dystrophic Epidermolysis Bullosa : Standard Dressing Versus Amniotic Membrane.
Brief Title: A Comparative Study of the Healing of Chronic Ulcers of Recessive Epidermolysis Bullosa : Dressing vs Amniotic Membrane
Acronym: MABUL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P130907 - 2014-001805-42
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Epidermolysis Bullosa Dystrophica, Recessive; Ulcer
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Ulcer | interventions — Biological Dressings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Dressing (Active Comparator): J0 to J42 : once a week, primary dressing with Mepitel®
  Interventions: Device: Amniotic Membrane
- Amniotic Membrane (Experimental): J0 to J42: once a week, Mepitel® and amniotic membrane (one or several depending on the graft size, so that the ulcer was completely covered with MAH). The last amniotic membrane is left in place.
  Interventions: Device: Amniotic Membrane

INTERVENTIONS:
Device: Amniotic Membrane

SUMMARY:
Skin wounds of Recessive Epidermolysis Bullosa Dystrophica (REBD) involve pain, superinfection, protein-losing, inflammation, and joint contractures are the bed of squamous cell carcinoma. There is no precise data on the kinetics of healing post-bullous erosions but clinical experience suggests that most epidermise in less than a month. Some, however, for unknown reasons, persist for several months. These chronic ulcers (UC), arbitrarily defined for this study as lasting more than three months are a source of major discomfort and could play a decisive role in the morbidity and mortality of the disease.

The aim of this study is to evaluate the efficacy of the amniotic membrane on the healing of chronic ulcers REBD on the percentage ulcerated surface re-epithelialised at 12 weeks (M3) from the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 years and 60
* REBD clinically evident with immunohistological confirmation and / or genetic
* REBD with at least two chronic ulcers (> 3 months) comparable
* Signing the informed consent of the patient and / or (children) of parents holding parental authority
* Affiliation to a social security scheme (beneficiary or legal)

Exclusion Criteria:

* Epidermoid carcinoma on the target or chronic ulcers
* Budding excessive requiring the application of a topical corticosteroid on the target or chronic ulcers
* Skin bacterial superinfection clinically overt requiring oral antibiotics
* Herpes simplex virus superinfection
* major evolutionary and malnutrition defined as a BMI <12 or more than 2 variant between screening and randomization OR a serum albumin <20 g / l or more ranging from 5 g / l between screening and randomization
* major and progressive anemia defined by a Hb <6 g / liter or variant more than 4 g / l between screening and randomization
* Life expectancy estimated at less than 3 months
* Pregnancy
* Inability to understand or observance of the rules of protocol
* Participation in another interventional therapeutic biomedical research whose treatment is not yet completed or the primary endpoint is not yet measured at the time of inclusion in Mabul

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of ulcerated area re-epithelialised | at 12 weeks from the start of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, Paris, France